CLINICAL TRIAL: NCT00779207
Title: Effect of Weight Loss and Exercise on Intrahepatic and Intramyocellular Fat in Obese Older Adults
Brief Title: Effect of Weight Loss and Exercise on Liver and Muscle Fat in Obese Elderly
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Washington Universtiy School of Medicine, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DK 37948A; R01AG025501 (NIH)
Record Dates: First submitted 2008-10-22; First posted 2008-10-24 (Estimated); Last update posted 2008-10-24 (Estimated); Status verified 2008-10

CONDITIONS: Obesity
Keywords: obesity; aging; exercise; diet; weight loss; physical function; Obesity in the Elderly
MeSH Terms: conditions — Obesity; Motor Activity; Weight Loss | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): weight loss
  Interventions: Behavioral: weight loss
- 2 (Experimental): Weight loss and exercise
  Interventions: Behavioral: weight loss and exercise

INTERVENTIONS:
Behavioral: weight loss and exercise — 10% weight loss through diet and exercise plus multicomponent exercise training three times a week
  Other Names: lifestyle modification
  Arms: 2
Behavioral: weight loss — 10 percent weight loss through diet and behavioral modification
  Other Names: lifestyle change
  Arms: 1

SUMMARY:
The purpose of this study is to determine the effect of weight loss and exercise on liver and muscle fat.

DETAILED DESCRIPTION:
Obesity causes serious medical complications and impairs quality of life. Moreover, both aging and obesity cause metabolic and physical dysfunction. The primary objectives of the proposed research are to evaluate the independent and combined effects of weight loss and exercise on Intrahepatic and Intramyocellular fat in obese elderly men and women. The central hypothesis is that in obese elderly subjects, weight loss will improve metabolic and physical function while the addition of exercise will not only augment improvement in these outcomes, but also attenuate the adverse effects of weight loss on bone and muscle masses. To test this hypothesis, 20 elderly (65-85 years old) obese men and women (body mass index [BMI] > 30 kg/m2) with physical frailty will be randomized to 2 treatment groups: 1)10% weight loss, 2) 10% weight loss plus exercise training.

ELIGIBILITY:
Inclusion Criteria:

* Obese (BMI 30 or greater)
* Elderly (age 65 years or older)

Exclusion Criteria:

* Major chronic disease or any condition that would interfere with exercise or dietary restriction, in which exercise or dietary restriction are contraindicated, or that would interfere with interpretation of results. Examples include cardiopulmonary disease, unstable disease, severe orthopedic or neuromuscular impairments, dementia, history of malignancy during the past 5 years

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-11; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Intrahepatic fat Intramyocellular fat | 6-month

SECONDARY OUTCOMES:
Insulin sensitivity Physical Function | 6-month

CONTACTS AND LOCATIONS:
Overall Officials: Dennis T Villareal, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Villareal DT, Banks M, Siener C, Sinacore DR, Klein S. Physical frailty and body composition in obese elderly men and women. Obes Res. 2004 Jun;12(6):913-20. doi: 10.1038/oby.2004.111. PMID 15229329